CLINICAL TRIAL: NCT01264055
Title: Cross-Sectional Characterization of Idiopathic Bronchiectasis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110046; 11-H-0046
Record Dates: First submitted 2010-12-18; First posted 2010-12-21 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-07-08

CONDITIONS: Infection; Bronchial Diseases; Respiratory Tract Diseases
Keywords: Rare Disease of Airways; Chronic Cough; Nontuberculous Mycobacteriam Infection; Natural History; Bronchiectasis; Idiopathic Bronchiectasis
MeSH Terms: conditions — Infections; Bronchial Diseases; Respiratory Tract Diseases; Chronic Cough; Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Adults with idiopathic bronchiectasis

SUMMARY:
Background:

- Bronchiectasis is a type of lung condition in which the lungs airways are abnormally stretched and widened. This stretching and widening makes it difficult for mucus and other substances to move out of the lungs, encouraging the growth of bacteria and leading to breathing problems or infection. Bronchiectasis can be caused by genetic disorders or diseases such as tuberculosis or rheumatoid arthritis. Researchers are interested in developing better ways to diagnose and treat a lung problem called idiopathic or unexplained bronchiectasis.

Objectives:

- To better describe the physical characteristics, radiographic patterns, and airway microbiology of unexplained bronchiectasis and to look for possible genetic links or risk factors.

Eligibility:

* Individuals at least 18 years of age who have a chronic cough and who have had a CT scan that has revealed signs of bronchiectasis.
* Current smokers or those who have smoked for at least 10 years, as well as individuals who have known causes of bronchiectasis or who have had organ transplants, are not eligible to participate.

Design:

* Participants will have one outpatient clinic visit for evaluation with a physical examination including detailed body size measurements and medical history and for collection of blood samples for routine lab tests and genetic analyses and a chest x-ray if no recent one is available.
* Participants will also have tests of lung function, and measurement of a gas called nitric oxide in the nose. Participants whose initial tests show abnormal results may also be asked to have a nasal scrape to collect cell samples and/or a skin sweat test to measure salt concentrations.
* Participants will also have a sputum specimen collected during the visit and will be asked to collect two additional early morning sputum samples and a mouth rinse at home within 2 weeks of the clinic visit, and mail the sample collection materials to the research team.

DETAILED DESCRIPTION:
The Genetic Disorders of Mucociliary Clearance Consortium (GDMCC) is comprised of 6 geographically-dispersed clinical research sites designed to study chronic disorders of the conducting airways associated with bronchiectasis. The first Clinical Center protocol (06-I-0217) focused on airway diseases with a known genetic etiology: primary ciliary dyskinesia (PCD), variant cystic fibrosis (vCF), and pseudohypoaldosteronism (PHA). This second GDMCC protocol will study adult patients with non-CF, idiopathic bronchiectasis, whose genetic etiologies are not known. Patients will receive the same level of rigorous testing that has allowed proper diagnosis of patients with PCD, vCF, and PHA.

Idiopathic bronchiectasis is reportedly more common in females with certain asthenic morphotypes and associated with environmental organisms, such as nontuberculous mycobacterium (NTM). Gender predilection due to referral bias is unclear. Other susceptibility factors predisposing to bronchiectasis or acquisition of NTM are also unclear.

The study will attempt to broaden the understanding of this disease by comparing gender-associated factors and NTM status. A relatively equal number of both females/males and NTM/non-NTM infected subjects will be accrued. Patients will be stratified by gender and by the presence/absence of respiratory infection with NTM. Approximately 300 people may be screened to find 260 eligible subjects since a small number (e.g., 40 patients) may be diagnosed with PCD, vCF, or other known etiology as an explanation for the bronchiectasis.

This single-visit protocol will use a systematic approach to characterize the clinical, morphological, radiological, and microbiological phenotypes of idiopathic bronchiectasis. Physical features, radiographic patterns, and associated lower airway microbial flora will be assessed. There is no natural history of disease course follow-up component to this protocol. The standard evaluation includes a quantitative assessment of body morphometrics, functional assessments of pulmonary physiology, nasal nitric oxide measurement with subsequent detailed assessment of ciliary structure and motility in selected patients, quantitative immunoglobulins levels to screen for humoral immune defects, and selected genetic analysis of candidate alleles, such as CFTR and A1AT.

Genotype/phenotype correlations will be researched and possibly defined. Careful evaluation and characterization of these phenotypes will guide the genetic characterization of idiopathic bronchiectasis, and likely lead to an improved diagnostic approach. Identification of disease causing genes may provide new therapeutic targets.

ELIGIBILITY:
* INCLUSION CRITERIA:

The criteria for participants to enter the study mandates that each patient have received a standard (current clinical practice) diagnostic evaluation that includes a CT scan of the chest to document bronchiectasis, prior to enrolling in the Consortium study. To enter this protocol, adults must have bronchiectasis and meet the following criteria:

1. Males or females, age greater than or equal to18 years
2. Chronic cough
3. An available CT of the chest (on a CD) that shows evidence of dilated airways fulfilling radiographic criteria for bronchiectasis in more than one lobe
4. Ability to provide informed consent, including HIPAA consent

EXCLUSION CRITERIA:

A participant should not be in the study if they have not had a standard clinical evaluation to rule out other potential causes of chronic sino-pulmonary disease.

1. Known diagnosis of cystic fibrosis with classic clinical presentation and elevated sweat chloride levels and/or two known disease-causing CFTR mutations
2. History of tuberculosis or other known explanation for bronchiectasis, such as alpha 1-antitrypsin deficiency (ZZ or ZS), confirmed or probable PCD, inflammatory bowel disease, rheumatoid arthritis, Sjogren s syndrome, allergic bronchopulmonary aspergillosis, or documented primary or acquired immunodeficiency
3. Current smoker or > 10 pack-year history of tobacco use
4. Prior solid organ transplant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with idiopathic bronchiectasis, with stratification by gender and by presence/absence of respiratory infection with nontuberculous mycobacteria (NTM)
Sampling Method: Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2011-04-26 (Actual)

PRIMARY OUTCOMES:
Clinical characteristics by gender and NTM | 30 years
  Clinical characteristics by gender and NTM status including body morphotypes, radiographic patterns, and respiratory flora

SECONDARY OUTCOMES:
Seek to define Genotype/phenotype | 30 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Lipton, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (6):
- United States (5):
  - Stanford Medical Center, Stanford, California
  - National Jewish Health, Denver, Colorado
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Washington University, St. Louis, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
- St. Michael's Hospital, Toronto, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wanner A, Salathe M, O'Riordan TG. Mucociliary clearance in the airways. Am J Respir Crit Care Med. 1996 Dec;154(6 Pt 1):1868-902. doi: 10.1164/ajrccm.154.6.8970383. No abstract available.
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-H-0046.html